CLINICAL TRIAL: NCT00600795
Title: Prognostic Value of Transforming Growth Factor-Beta 1 in Normal Pressure Hydrocephalus
Status: Completed | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 070875
Record Dates: First submitted 2008-01-07; First posted 2008-01-25 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-03

CONDITIONS: Normal Pressure Hydrocephalus
Keywords: NPH; TGF-beta
MeSH Terms: conditions — Hydrocephalus, Normal Pressure; Camurati-Engelmann Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — CSF
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- A: Patients diagnosed with Normal Pressure Hydrocephalus
  Interventions: Other: CSF collection

INTERVENTIONS:
Other: CSF collection — CSF collection at time of VPS insertion

SUMMARY:
Correlation of cerebrospinal fluid levels of transforming growth factor beta-1 with functional improvements after insertion of ventriculoperitoneal shunt for normal pressure hydrocephalus

DETAILED DESCRIPTION:
The goal of this research is to investigate a potential CSF biomarker of NPH as a new tool for both the diagnosis of NPH and prognosis of VPS placement. Transforming growth factor-b1 (TGF-b1) is a signaling molecule involved in three fundamental activities; suppression of cell proliferation, immunosuppression, and deposition of extracellular matrix through promotion of synthesis and inhibition of degradation.8 Previously, TGF-b1 had been implicated in the development of communicating hydrocephalus secondary to pre-term infant intraventricular hemorrhage9 and adult aneurysmal sub-arachnoid hemorrhage.10, 11 Recently, an investigation demonstrated elevated levels of TGF-b1 in patients with shunt-responsive NPH compared to non-NPH patients.12

The specific aims of this research proposal are to:

1. Correlate CSF levels of TGF-b1 with the clinical response of patients diagnosed with NPH to VPS placement.
2. Correlate CSF levels of TGF-b1 with optimal VPS pressure settings.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Normal Pressure Hydrocephalus

Exclusion Criteria:

* Patients not diagnosed with Normal Pressure Hydrocephalus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinic and neurology clinic
Sampling Method: Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2008-01; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
TGF beta-1 levels | Time of Surgery
Mini-mental status exam | Pre-operative, 3 and 12 months post-operatively
Modified barthel index | Pre-operative, 3 and 12 months post-operatively
Tinetti mobility assessment | Pre-operative, 3 and 12 months post-operatively

SECONDARY OUTCOMES:
Programmable shunt setting | Pre-operative, 3 and 12 months post-operatively

CONTACTS AND LOCATIONS:
Overall Officials: Noel Tulipan, M.D., Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States